CLINICAL TRIAL: NCT04820998
Title: Living in a Precarious Situation With an Autistic Child: What Are the Issues at Stake for Support in Care: Qualitative Study - Monocentric Study
Brief Title: Living in a Precarious Situation With an Autistic Child: What Are the Issues at Stake for Support in Care
Acronym: HaSPrEA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH029
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Autistic Disorder
Keywords: precarious; support; care; professional interview; family interview
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Families — Families's interviews about their precarious situation of living and the consequences on their autistic child care
Other: professionals — Interviews so as to know how the specifics of precarious situations are identified and taken into account by the professionals

SUMMARY:
Study the specificities of families in a precarious situation with a child with autism spectrum disorders (ASD) in terms of housing, in order to better support them in the various social spaces and improve collaboration between professionals and parents

DETAILED DESCRIPTION:
Identify the living conditions related to the housing of children with autism spectrum disorders (ASD) treated at the Léo Kanner Center (CLK), psychopathology department of the Saint-Étienne University Hospital. The aim is to describe through the trajectories of children with ASD and their families, their living conditions, and through interviews with professionals who support them, how the specificities related to precarious situations are identified and taken into account.

A qualitative survey, carried out by sociological interviews with families whose children are followed at the Léo Kanner Center (CLK) and the professionals who care for them, would make it possible to collect data on the development of a young child with autism in his home and more generally in his habitat.

The purpose of this study is to study the specificities of families in a precarious situation with a child with autism spectrum disorders (ASD) in terms of housing, in order to better support them in different social spaces and improve collaboration between professionals and parents. The project aims to bring children with autism spectrum disorders (ASD) into a dynamic of access to human rights. He suggests three levers to achieve this: rely on a precise inventory of needs; work towards a transformation of representations; streamline access to healthcare and common law services.

ELIGIBILITY:
Inclusion Criteria:

* Families having their child followed in the child psychiatry service of the Léo Kanner Center (CLK),
* Children followed for Autism Spectrum Disorders (ASD),
* Families who received informed information about the study and who co-signed a consent to participate in the study with the investigator.

Exclusion Criteria:

* Opinion of the child's referring physician contraindicating inclusion
* Refusal of one of the legal guardians to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children followed for Autism Spectrum Disorders (ASD)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
living conditions of children with Autism Spectrum Disorders (ASD) | hours 2
  To identify the living conditions related to the housing of children with Autism Spectrum Disorders (ASD) who are cared for at the Léo Kanner Center (CLK), psychopathology department of the University Hospital of Saint-Etienne.

SECONDARY OUTCOMES:
Precarity | hours 2
  Families's interviews about their precarious situation of living and the consequences on their autistic child care

OTHER OUTCOMES:
Professionals | hours 2
  Interviews so as to know how the specifics of precarious situations are identified and taken into account by the professionals

CONTACTS AND LOCATIONS:
Overall Officials: VALERIE ROUSSELON-CHARLES, MD, Principal Investigator — CHU ST ETIENNE FRANCE
Locations (1):
- Chu St Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No